CLINICAL TRIAL: NCT04706143
Title: T Cell, Antibody and Cytokine Responses to Single and Double Doses of COVID-19 Vaccines in Egyptians
Brief Title: Immunologic Responses to Single and Double Doses of COVID-19 Vaccines in Egyptians
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU21
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Vaccines
Keywords: COVID-19; Safety; Efficacy; T cell responses; Cytokine responses; Antibody responses
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccined group by live attenuated or viral vector or mRNA vaccine: Adults between 25-65 years old
  Interventions: Biological: COVID-19 Vaccines

INTERVENTIONS:
Biological: COVID-19 Vaccines — different available vaccines: live inactivated, mRNA and viral vector vaccines

SUMMARY:
The recent Coronavirus Disease 2019 (COVID-19), has caused a global pandemic, and development of safe, effective vaccines is mandatory to return back to pre pandemic life. Many vaccines have been developed and requested by the authorities after the emergency license issued. The main mechanism of protection is through humoral and cell-mediated immune responses that might reduce the potential for disease development or severity. Cytotoxic T cells clear virus-infected host cells and contribute to control of infection. Preliminary data are now available indicating safty and effecacy of different vaccines . The vaccines were tolerated, with induction of neutralizing antibodies and antigen-specific T cells against the SARS-CoV-2 spike protein. The aim of this work is to evaluate the immune responses in adults, aged 25-65 years, up to 8 weeks after vaccination with a single and double doses live inactivated (Sinopharm), mRNA (Pfizer/ Biontech) and viral vector (Oxford/AZ- ChAdOx1 nCoV-19) vaccines. The Th1- response ( interferon-γ and tumor necrosis factor-α cytokine secretion by CD4+ T cells) and antibody production predominantly of IgG1 and IgG3 subclasses as well as CD8+ T cells mono, polyfunctional and cytotoxic phenotypes, will be also measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults receiving COVID-19 vaccines

Exclusion Criteria:

* any contraindication of each COVID-19 vaccine as listed by WHO

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults aged from 25-65 years old non immune-compromised or immune suppressed receiving COVID-19 vaccines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
measure immune cell activation induced by the vaccine | 8 weeks
  estimate number of lymphocytes, T cells, Natural killer cells and B cells
measure antibody response to vaccines | 8 weeks
  evaluation of IgG and IgM levels, mg/dl
measure the cytokine response to different vaccines | 8 weeks
  level of IL-1, IL-2, TNF-alpha, IFN- gamma, My/dl

IPD SHARING:
Plan to Share IPD: Yes
On request